CLINICAL TRIAL: NCT02653716
Title: BeST?- The Best Services Trial (BeST?): Effectiveness and Cost-effectiveness of the New Orleans Intervention Model for Infant Mental Health
Brief Title: Effectiveness and Cost-effectiveness of the New Orleans Intervention Model for Infant Mental Health
Acronym: BeST?-
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helen Minnis (Other)
Collaborators: University of Glasgow (Other); National Institute for Health Research, United Kingdom (Other Government); King's College London (Other); Glasgow City Council Social Work (Unknown); National Society for the Prevention of Cruelty to Children (Other); NHS Greater Glasgow and Clyde (Other); University of Aberdeen (Other)
Responsible Party: Sponsor-Investigator, Helen Minnis, Professor of Child and Adolescent Psychiatry, University of Glasgow
Organization: University of Glasgow (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: GN14CO183
Record Dates: First submitted 2015-12-23; First posted 2016-01-12 (Estimated); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Maltreatment; Mental Health
Keywords: New Orleans Intervention Model; Case Management; Maltreatment; Child
MeSH Terms: conditions — Psychological Well-Being | interventions — Case Management

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case Management (Active Comparator): CM
  Interventions: Behavioral: Case Management
- New Orleans Intervention Model (Experimental): NIM
  Interventions: Behavioral: New Orleans Intervention Method

INTERVENTIONS:
Behavioral: New Orleans Intervention Method — An attachment based assessment, then a tailored intervention aimed at maximising the chances of the maltreated child being returned to the birth family
  Arms: New Orleans Intervention Model
Behavioral: Case Management — A social work assessment of family functioning that makes future recommendations regarding the future placement of a maltreated child.
  Arms: Case Management

SUMMARY:
To evaluate the clinical and cost-effectiveness of the New Orleans Intervention Method (NIM) in relation to an enhanced services as usual model, Case Management (CM), for the management of maltreated infants and young children entering care in the United Kingdom (UK) .

DETAILED DESCRIPTION:
Children who have experienced abuse and neglect are at increased risk of mental and physical health problems throughout life. This places an enormous burden on individuals, families and society. Regardless of the severity of this abuse and neglect, these negative effects can largely be reversed if children are placed in secure, loving homes early enough in life. Placing children in nurturing foster placements can help them recover rapidly, but it is not known whether it is better for children's long term development to place them with substitute (foster or adoptive) families or return them to birth or extended families. Efforts to improve the mental health of maltreated children in birth families or foster placements have had mixed success and researchers have recommended that far more intensive approaches are required.

The investigators have carried out careful exploratory research, in Glasgow, on an intensive approach, which was developed in the United States. This is was investigators have called this the New Orleans Intervention Model (NIM). NIM offers families who have a child who enters care due to abuse or neglect a structured assessment of family relationships followed by an intensive treatment that aims to improve family functioning and child mental health. If adequate change is achieved a recommendation is made for the child to return home but, if not, the recommendation is for adoption. Preliminary research from the US suggests that NIM might reduce future maltreatment of the child and other children in the family, and improve mental health in middle childhood.

The investigators are currently conducting a study in which, since December 2011, has recruited around two-thirds of all maltreated children aged 0 to 5 years coming into an episode of care in Glasgow. Half of the families who are taking part receive NIM, which is delivered by a multidisciplinary team comprising health and social care professionals. The remaining half of families will receive usual services, which is delivered by social workers. Preliminary findings suggest that NIM is acceptable to parents, foster carers, social workers and legal professionals. Investigators added an additional site, London, as there is a need to test whether NIM is effective, in terms of both clinical outcomes and cost, in the different legal systems across England and Scotland. The plan is to launch NIM teams at these sites in 2016.

The Investigators, therefore, propose a study of NIM involving a continuation of our current Glasgow work and including 1-2 additional sites. This will involve approximately 500 children (396 families) in total across the sites, including those recruited in our current Glasgow internal pilot study. This will determine whether or not NIM is effective in the UK and to follow up Glasgow children for five years to examine longer term effects on mental health.

ELIGIBILITY:
Inclusion Criteria:

* Family with a child aged 0-60 months who enters care in the recruiting sites for reasons associated with maltreatment during the study recruitment period.

Exclusion Criteria:

* Families will be excluded from the trial if the parent(s) is unavailable to take part in intervention (e.g. because of death, unknown whereabouts or long term imprisonment).

Ages: 0 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 384 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
Child mental health measured by the Total Difficulties scale of the Strengths and Difficulties Questionnaire to establish if NIM in relation to CM is effective in improving child mental health as evidenced by reduced scores. | 30 months after the last participant has been recruited
  A brief behavioural screening questionnaire for 2-17 year-olds completed by the primary caregiver with 25 items in 5 subscales: emotional symptoms; conduct problems; hyperactivity/inattention; peer relationship problems and prosocial behaviour

SECONDARY OUTCOMES:
Improvement in the relationship between the primary caregiver and the maltreated child as evidenced by increased scores on the Parent-Infant Global Assessment Scale (PIR-GAS)" | 30 months after the last participant has been recruited
Quality of life by reviewing the PedsQL - a measure of child quality of life to look at Quality Adjusted Life Years (QALYs) | 30 months after the last participant has been recruited

CONTACTS AND LOCATIONS:
Overall Officials: Helen Minnis, Principal Investigator — University of Glasgow
Locations (2):
- United Kingdom (2):
  - University of Glasgow, Glasgow
  - Kings College London, London

REFERENCES:
- [Derived] Crawford K, Young R, Wilson P, Deidda M, Forde M, Millar S, McConnachie A, Boyd K, McIntosh E, Ougrin D, Henderson M, Gillberg C, Kainth G, Turner F, Sonuga-Barke EJS, Fitzpatrick B, Minnis H. Infant mental health services for birth and foster families of maltreated pre-school children in foster care (BeST?): a cluster-randomized phase 3 clinical effectiveness trial. Nat Med. 2025 May;31(5):1617-1625. doi: 10.1038/s41591-025-03534-9. Epub 2025 May 1. PMID 40312587
- [Derived] Deidda M, Boyd KA, Minnis H, Donaldson J, Brown K, Boyer NRS, McIntosh E; BeST study team. Protocol for the economic evaluation of a complex intervention to improve the mental health of maltreated infants and children in foster care in the UK (The BeST? services trial). BMJ Open. 2018 Mar 14;8(3):e020066. doi: 10.1136/bmjopen-2017-020066. PMID 29540420